CLINICAL TRIAL: NCT05767606
Title: Safety and Immunogenicity of Concomitant Administration of the Novavax Vaccine and a 20-valent Pneumococcal Conjugate Vaccine in Adults Aged ≥60 Years: a Four-arm, Double-blind, Non-inferiority Trial
Brief Title: Concomitant Administration of the Novavax Vaccine and a 20-valent Pneumococcal Conjugate Vaccine in Adults Aged ≥60 Years
Acronym: NVX_PCV20
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Markus Zeitlinger, Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NVX_PCV20_V2.1
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Pneumococcal Infections
MeSH Terms: conditions — COVID-19; Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- NVX arm (Active Comparator): NVX plus placebo
  Interventions: Biological: NVX
- PCV20 arm (Active Comparator): PCV20 (Apexxnar®) plus placebo
  Interventions: Biological: PCV20
- Combination arm (Experimental): NVX plus PCV20
  Interventions: Biological: NVX; Biological: PCV20
- Placebo arm (Placebo Comparator): Placebo (normal saline) plus placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NVX — Administration of NVX
  Arms: Combination arm; NVX arm
Biological: PCV20 — Administration of PCV20
  Arms: Combination arm; PCV20 arm
Biological: Placebo — No intervention
  Arms: Placebo arm

SUMMARY:
Vaccination is a key strategy for preventing respiratory illnesses. Pneumococcal vaccination is recommended for all adults aged over 60 or 65 years (depending local guidelines) who have never received a pneumococcal vaccine or whose previous vaccination history is unknown. Given their wide application, co-administration of pneumococcal and Covid-19 vaccines may support broad population-wide coverage. However, it is unclear whether the co-administration of the Novavax (NVX) vaccine and a 20-valent pneumococcal conjugate vaccine (PCV20) results in lower immunogenicity than the administration of either alone.

The investigators will thus conduct a 4-four arm study with the following treatments: NVX plus placebo (NVX arm), PCV20 plus placebo group (PCV20 arm), NVX plus PCV20 (Combination arm), and placebo plus placebo group (Placebo arm). Vaccines and/or placebo will be administered as single doses, given as intramuscular injections on Day 1 (one in each shoulder). Subjects will be randomly assigned to one of the four arms.

The outcome will be the antibody levels after 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60 years or older
* Males and females
* Able and willing (in the investigator's opinion) to comply with all study requirements.
* Participants, who already received three Covid-19 vaccines, of which the third was a mRNA vaccine (BNT162b2 or mRNA-1273) and at least 16 weeks ago
* Only applicable for women: last menstrual bleeding more than one year ago

Exclusion Criteria:

* Use of immunosuppressants
* Congenital or acquired immunodeficiency (eg, history of HIV infection, hematological disease, current malignancy, or others)
* Chronic condition that may significantly interfere with the immune response in the opinion of the investigator
* History of Covid-19 within 16 weeks before study vaccination
* Previous pneumococcal vaccination
* Contraindication against any ingredient of the NVX or the PCV20 vaccine

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | Day 28
  Antibody levels

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jorda A, Prager M, Pracher L, Haselwanter P, Jackwerth M, Al Jalali V, Yildiz E, Leutzendorff A, Weber M, Yourieva S, Kammerer P, Pecho T, Decaminada A, Ederer L, Wiedermann U, Weseslindtner L, Redlberger-Fritz M, Bergmann F, Zeitlinger M. Immunogenicity, safety, and reactogenicity of concomitant administration of the novavax vaccine against Omicron XBB.1.5 (NVX-CoV2601) and a 20-valent pneumococcal conjugate vaccine in adults aged >/=60 years: A randomised, double-blind, placebo-controlled, non-inferiority trial. J Infect. 2025 Feb;90(2):106405. doi: 10.1016/j.jinf.2024.106405. Epub 2025 Jan 3. PMID 39756693